CLINICAL TRIAL: NCT04704362
Title: Ensuring Quality in Psychological Support
Acronym: EQUIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: World Health Organization (Other); The Center for Victims of Torture, United States (Other); University of Washington (Other); University of Nairobi (Other); War Child Holland (Unknown); Socios En Salud Sucursal, Peru (Other); University of South Florida (Other); HealthRight International (Unknown); Johns Hopkins University (Other); Centre for Infectious Disease Research in Zambia (Other); The University of New South Wales (Other)
Responsible Party: Principal Investigator, Brandon A Kohrt, MD, PhD, Associate Professor, George Washington University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCR191797
Record Dates: First submitted 2020-07-29; First posted 2021-01-11 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Psychological Distress; Depression
Keywords: Training; Competency; Mental health; Psychological treatment
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Organization and Administration

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled trial comparing training and supervision as usual with training and supervision using a competency-based approach.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trainees and their patients will not be told which arm the trainee was in. Outcome assessors will also be blinded to arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training and Supervision as Usual (Active Comparator): Non-specialists are trained in a psychological intervention under standard conditions. No feedback from competency-based evaluations is provided to modify the training or supervision curriculum.
  Interventions: Behavioral: Standard Training and Supervision
- Competency-based Training and Supervision (Experimental): Non-specialists are trained and supervised in a competency-based approach in which trainers and/or supervisors are provided with the competency scores of trainees in order to modify the training and supervision content and approach as needed.
  Interventions: Behavioral: Ensuring Quality in Psychological Support

INTERVENTIONS:
Behavioral: Ensuring Quality in Psychological Support — Trainees are evaluated with the Enhancing Assessment of Common Therapeutic factors structured role play tool and the results are shared with trainers and/or supervisors to modify training based on strengths and weakness on the competency scores.
  Arms: Competency-based Training and Supervision
Behavioral: Standard Training and Supervision — Trainees are trained using a manual for non-specialist-delivered psychological interventions.
  Arms: Training and Supervision as Usual

SUMMARY:
The goal of this project is to test tools that will be part of a platform for training and supervision of mental health and psychosocial support helpers, including providers without specialized training in mental health. This platform, entitled Ensuring Quality in Psychological Support, is an online resource being developed to include: materials for evaluating core and specific competencies, training on core competencies, implementation guidance to conduct competency-based training. The Ensuring Quality in Psychological Support platform is designed to aid trainers and supervisors working with providers being trained to deliver World Health Organization and non-World Health Organization low-intensity psychological interventions. The research will address two study objectives: Objective 1. Determine feasibility, acceptability, and perceived utility of the Ensuring Quality in Psychological Support platform; Objective 2. Evaluate the reliability, validity, and sensitivity to change of Ensuring Quality in Psychological Support competency assessment tools. To maximize generalizability of findings, Ensuring Quality in Psychological Support will be evaluated in seven countries: Ethiopia, Kenya, Lebanon, Peru, Uganda, Zambia and Jordan. The sites are varied by types of psychological intervention, beneficiaries, experience of trainers, and background of trainees. In each site, trainers will train non-specialist providers on a low-intensity psychological intervention.

DETAILED DESCRIPTION:
There is increasing evidence that non-specialist or minimally trained mental health providers can effectively provide support and deliver psychosocial support and low-intensity psychological interventions for common mental disorders and substance use disorders in low resource settings. Psychological treatments delivered by non-specialists in low-resource settings have effectiveness comparable to high-income country studies of specialist interventions.

Low intensity interventions refer to interventions that do not rely on specialists and are modified, brief evidence-based therapies including guide self-help and e-mental health. The World Health Organization identifies such interventions as being: brief, basic, non-specialist-delivered versions of existing evidence-based psychological treatments (e.g., basic versions of cognitive-behavioral therapy, interpersonal therapy); and may include self-help materials (e.g., self-help books, audiovisual materials, and online or app-based self-help interventions); individual or group programs, and designed to be age-appropriate (i.e., delivered differently for children and adults). Moreover, low intensity interventions are particularly well suited to communities affected by adversity, as they use fewer resources which make them more scalable.

Psychosocial refers to interventions that are designed to address the psychological effects of conflict [or adversity], including the effects on behavior, emotion, thoughts, memory and functioning, and social effects, including changes in relationships, social support and economic status. The term psychosocial emphasizes, the close connection between psychological aspects of experience and wider social aspects of experience, inclusive of human capacity, social ecology, and culture and values. For the purpose of this study, low intensity psychological and psychosocial interventions were selected using the criteria above, and ensuring the interventions are freely accessible to the public.

To assure success of such interventions outside the context of resource-intensive research trials, it is crucial to develop training and supervision programs that produce competent providers of psychological and psychosocial support interventions. A necessary element to achieve this goal is development of standardized tools and procedures to assess the competency of those trained to deliver them; while ensuring competency assessment results are easily understandable to trainers and supervisors so that they can remediate areas of low competency.

In the context of psychological and psychosocial interventions, competency refers the extent to which a therapist [including non-specialists] has the knowledge and skill required to deliver a treatment to the standard needed for it to achieve its expected effects. Competency is typically assessed through structured role-plays in which trained standardized [mock] clients elicit trainee's ability to perform the key skills of an intervention. Role-plays such as this are commonly used in health professional training and evaluation in the form of observed structured clinical evaluations with simulated patients. The Ensuring Quality in Psychological Support initiative was developed out of need to have easily implementable competency evaluation tools and remediation training materials that can be used with specialists and non-specialists in diverse global settings. To supplement the platform, Ensuring Quality in Psychological Support will also include various implementation, trainer and training resources and guidance.

The need for these competency assessment tools and training materials was identified in May 2018, during a Theory of Change Workshop conducted by the World Health Organization Ensuring Quality in Psychological Support team with frontline psychological service practitioners, clinicians, non-governmental organization training and supervision staff, and researchers. The four key elements of the platform will be (a) competency tools for evaluation of non-specific (core competencies or common factors) and specific practice elements (or treatment specific factors); (b) role-play vignettes for conducting competency evaluations; (c) instructional materials on how to conduct competency evaluations (training standardized clients, establishing inter-rater reliability when conducting competency evaluations, using rating tools, interpreting results); and (d) instructional materials on how to integrate competency evaluations into trainings and supervision (giving feedback to participants, modifying training programs, feedback to trainers and supervisors) including core competency training and remediation materials.

Study Goals and Objectives:

The goal of the study is to inform development of the Ensuring Quality in Psychological Support platform and its tools, ensuring feasibility, acceptability, utility, reliability, and validity to support the provision of quality psychological support.

Study Objectives

1. Determine the feasibility, acceptability, and perceived utility, of the Ensuring Quality in Psychological Support platform to facilitate assessment of competency and employ competency assessment results and remediation training materials to support training and supervision of non-specialists on low-intensity psychological interventions.
2. Evaluate the reliability, validity, and sensitivity to change of Ensuring Quality in Psychological Support competency assessment tools based on inter-rater reliability of the tools within and between sites, ability to detect changes in competency over the course of training and supervision, and association with trainer ratings, as well as service delivery metrics and client outcomes across different psychological interventions and implementation sites.

ELIGIBILITY:
Inclusion Criteria:

* Trainees: Non-specialist in mental health and psychosocial support
* Clients: Site-specific level of distress to determine psychological intervention participation

Exclusion Criteria:

* Trainees: Unable to comprehend language that training and supervision will be conducted in
* Clients: Serious mental illness, developmental disability

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Trainee - Enhancing Assessment of Common Therapeutic factors; Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors" | Post-intensive supervision (approximately 1 month post-training)
  15-item objective structured clinical examination using a role play, minimum value = 15, maximum value = 60, higher score means greater competency

SECONDARY OUTCOMES:
Trainee - Enhancing Assessment of Common Therapeutic factors; Unabbreviated scale title: "Enhancing Assessment of Common Therapeutic Factors" | immediately after the manualized psychological treatment training
  15-item objective structured clinical examination using a role play, minimum value = 15, maximum value = 60, higher score means greater competency
Trainee - Trainer Subjective Rating of Competency; unabbrievated scale title "Trainer Subjective Rating of Competency" | immediately after the manualized psychological treatment training
  Trainer's subjective competency rating of trainee on a scale from 1 to 4, with higher scores reflecting greater competency.
Trainer's subjective competency rating of trainee on a scale from 1 to 4, with higher scores reflecting greater competency. | Post-intensive supervision (approximately 1 month post-training)
  Trainer's subjective competency rating of trainee on a scale from 1 to 4, with higher scores reflecting greater competency.
Trainee - Equip-Treatment-specific competencies; unabbreviated title "Ensuring Quality in Psychological Support Treatment Specific Competency" | Immediate post-training (last day of training on manualized intervention)
  Site specific measure of trainee's competencies in manualized psychological intervention delivered by non-specialists; mean scores range from 1=potentially harmful, 2=some basic skills; 3=all basic skills; 4=advanced skills; higher score is more competency
Trainee - Equip-Treatment-specific competencies; unabbreviated title "Ensuring Quality in Psychological Support Treatment Specific Competency" | Post-intensive supervision (approximately 1 month post-training)
  Site specific measure of trainee's competencies in manualized psychological intervention delivered by non-specialists; mean scores range from 1=potentially harmful, 2=some basic skills; 3=all basic skills; 4=advanced skills; higher score is more competency
Client - mental health outcome, for example, Patient Health Questionnaire; unabbreviated title "Patient Health Questionnaire" | Immediately after completion of the manualized psychological treatment
  Site specific mental health outcome measure of client; higher scores reflect greater psychological distress; for example, Patient Health questionnaire range from 0 to 27; greater score is more symptoms.
Client - functioning outcome, for example, unabbreviated title: "World Health Organization Disability Assessment Schedule" | Immediately after completion of the manualized psychological treatment
  Site specific client functional impairment measure; higher scores reflect greater functional impairment; for example, World Health Organization Disability Assessment Schedule score range from 0 to 60; greater score is more impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Schafer, PhD, Principal Investigator — World Health Organization
Locations (7):
- Center for Victims of Torture, Addis Ababa, Ethiopia
- Institute for Family Health, Amman, Jordan
- University of Nairobi, Nairobi, Kenya
- War Child Holland, Beirut, Lebanon
- Socios en Salud Sucursal Peru, Lince, Peru
- HealthRight International Uganda, Kampala, Uganda
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared after completion of primary outcome publications from all sites.
Supporting Information: ICF
Time Frame: Individual participant data will be shared after completion of primary outcome publications from all sites.
Access Criteria: Contact principal investigator.